CLINICAL TRIAL: NCT05893940
Title: Low-Intensity Mechanical Stimulation for Hematologic Malignancy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I-3434822
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIMS vibration Therapy, DEXA Scan - Cohort 1 (Experimental): Patients undergo LIMS vibration therapy over 10 minutes on study. Patients also undergo DEXA scan at follow up and may optionally undergo blood sample collection and questionnaire at baseline and follow up
  Interventions: Procedure: Low Intensity Vibration Therapy; Procedure: Dual X-ray Absorptiometry; Procedure: Biospecimen Collection
- LIMS vibration therapy - Cohort II (Experimental): Patients undergo LIMS vibration therapy over 10-minutes BID for 14 days on study. Patients also undergo blood sample collection throughout the trial.
  Interventions: Procedure: Low Intensity Vibration Therapy; Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Low Intensity Vibration Therapy — Undergo LIMS vibration therapy
  Other Names: LIV; Low Intensity Virbration
Procedure: Dual X-ray Absorptiometry — Undergo DEXA scan
  Other Names: BMD scan; bone mineral density scan; DEXA
  Arms: LIMS vibration Therapy, DEXA Scan - Cohort 1
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This clinical trial tests the effect of low-intensity mechanical stimulation (LIMS) vibration therapy in patients with hematologic malignancies. Patients with hematologic malignancies often undergo a blood and/or bone marrow transplant (hematopoietic cell transplantation [HCT]) or cellular therapy. The LIMS board delivers vibrations through the bones that may stimulate bone growth and may also increase muscle activity and strength and may also increase T-cell activation in patients planning to undergo cellular therapy. LIMS vibration therapy may stop or reverse BMD loss and/or improve the development of T-cells in the body in patients with hematologic malignancies who are undergoing or may plan to undergo HCT or cellular therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of delivering a low-intensity mechanical stimulation (LIMS) program immediately following hematopoietic cell transplantation (HCT). COHORT 1 II. II. Evaluate chimeric antigen receptors (CAR) T-cell product efficacy of Non-Hodgkin lymphoma (NHL) patients undergoing LIMS in comparison to patients not treated with LIMS. COHORT II

SECONDARY OBJECTIVE:

I. Determine the effect size of a LIMS program on bone marrow density (BMD) post-HCT.

COHORT 1 II. Evaluate the manufacturing parameters (product viability, total cell dose, transduction efficiency, time to produce the CAR T-cell product) pre- and post-LIMS. COHORT II

OUTLINE:

Patients are assigned to 1 of 2 cohorts.

COHORT 1 - Patients undergo LIMS vibration therapy over 10-minutes once a day on study. Treatment begins day -8 to -1 during admission for HCT and until day 180 using the LIMS board at home. Patients also undergo dual x-ray absorptiometry (DEXA) scan at follow up and may optionally undergo blood sample collection at baseline and follow up.

COHORT II: Patients undergo LIMS vibration therapy over 10-minutes twice daily (BID) for 14 days on study. Patients also undergo blood sample collection throughout the trial

ELIGIBILITY:
Inclusion Criteria:

* COHORT I: Meet eligibility criteria for first autologous or allogeneic HCT (patients with preexisting osteoporosis are eligible)
* COHORT I: Scheduled to undergo an autologous or allogeneic HCT
* COHORT 1: >= 18 years of age
* COHORT 1: Patient must understand the investigational nature of this study and sign an institutional review board approved written informed consent form prior to receiving any study related procedure

  - COHORT II: ≥ 18 years of age
* COHORT II: Diagnosis of non-Hodgkin lymphoma (specifically diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, chronic lymphocytic leukemia; patients with preexisting osteoporosis are eligible)
* COHORT II: Patient must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

COHORT 1:

* Any prior allogeneic HCT
* Any prior autologous HCT for those patients who have a planned auto HCT
* Pre-transplant weight >= 275 lbs. (max weight for the board)
* Body mass index (BMI) < 18 kg/m^2
* Recipient of cord blood transplant
* Multiple myeloma or amyloidosis diagnosis
* History of a central nervous system (CNS) hemorrhage < 60 days
* History of any aneurysm (cerebral, aortic, etc.)
* A recent pulmonary embolism or deep vein thrombosis
* A cardiac pacemaker
* Prior history of non-traumatic (spontaneous) fracture
* Total joint replacement (any joint)
* History of kidney stones or gall stones within the last 2 years unless a cholecystectomy was performed
* Any prosthetic lower extremity or limb
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study intervention

COHORTII:

* Planned CAR T-cell therapy within the next 2 months
* Prior CAR T-cell therapy
* Active treatment within the last 60 days
* Pre-transplant weight ≥ 275 lbs. (max weight for the board)
* BMI < 18 kg/m^2
* History of a CNS hemorrhage < 60 days
* History of any aneurysm (cerebral, aortic, etc.)
* A recent pulmonary embolism or deep vein thrombosis
* A cardiac pacemaker
* Recent history (< 60 days) of non-traumatic (spontaneous) fracture
* Recent surgery (< 60 days)
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
time spent on LIMS - Cohort I | Up to 120 days post hematopoietic cell transplantation (HCT)
  Will assess how much time and days use throughout study period
Chimeric antigen receptor (CAR) T-cell product efficacy - Cohort II | up to 120 days post hematopoietic cell transplantation
  Blood samples will be collected for CAR-T cell efficacy before and after LIMS sessions

SECONDARY OUTCOMES:
Change in lumbar spine bone mineral density (BMD) - Cohort 1 | Up to 120 days post - HCT
  dual x-ray absorptiometry (DEXA) scans conducted as standard of care. BMD pre-HCT and post-HCT of patients who received LIMS compared to those who did not. A Linear regression used to compare the changes.
Change in femur BMD - Cohort 1 | UP to 120 days post - HCT
  Assessed using DEXA scans conducted as standard of care. BMD pre-HCT and post-HCT of patients who received LIMS will be compared to those who did not. A linear regression used to compare the changes.
Barriers to LIMS- Cohort 1 | Up to 120 post -HCT
  Reasons why LIMS was not used
Change in patient reported outcomes - Cohort 1 | Pre HCT and at time of second DEXA: day +80
  Short form 36 will be used to assess physical activities - comprising of 36 questions with ranges from 0 (worst) to 100 (Best)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Herr, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP